CLINICAL TRIAL: NCT07063706
Title: Impact of Pharmaceutical Care on Patients Using Capecitabine: a Multicenter Randomized Clinical Trial
Brief Title: Pharmaceutical Care for Patients Using Capecitabine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Farmácia (Other)
Collaborators: Universidade Federal Fluminense (Other); Instituto Nacional de Cancer, Brazil (Other Government); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5.204.291; 5.313.716 (Other: INSTITUTO NACIONAL DE CANCER); 5.855.089 (Other: UNIVERSIDADE FEDERAL DO RIO DE JANEIRO)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cancer Colorectal; Cancer Gi; Capecitabine; Pharmaceutical Services; Adverse Drug Reaction (ADR)
Keywords: capecitabine; pharmaceutical services; quality of life; adverse effects
MeSH Terms: conditions — Colonic Neoplasms; Gastrointestinal Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: Participants in the control group received pharmaceutical guidance at the time of dispensing capecitabine and participants in the intervention group received pharmaceutical care through consultations carried out on the dates scheduled for collection of capecitabine at the pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group received pharmaceutical guidance at the time of dispensing capecitabine.
- Pharmaceutical care (Active Comparator): Participants in the intervention group received pharmaceutical care.
  Interventions: Other: Pharmaceutical Care

INTERVENTIONS:
Other: Pharmaceutical Care — Participants in the intervention group received pharmaceutical care
  Arms: Pharmaceutical care

SUMMARY:
This is a longitudinal, prospective and intervention study, which will be carried out with patients undergoing treatment with capecitabine, where the impact of pharmaceutical care will be evaluated.

DETAILED DESCRIPTION:
Pharmaceutical care (PC) is a professional service in which the pharmacist, actively and in direct interaction with the patient, seeks to achieve concrete health results through the use of medications that improve their quality of life, considering their socioeconomic and cultural context. Through the practice of PC, it becomes possible to detect drug-related problems (DRPs), in addition to the possibility of preventing and resolving negative outcomes associated with the drug (NMR). With recent advances in cancer treatment, the increasing use of oral antineoplastic agents has accelerated. Despite the advantages involved in the use of oral chemotherapy compared to intravenous chemotherapy, there are associated risks that can compromise patient safety and the effectiveness of anticancer therapy. PC as a strategy to ensure and promote the safe and rational use of oral antineoplastics has been increasingly used in the care of cancer patients.

This is a longitudinal, prospective, interventional study that will be conducted with patients undergoing treatment with capecitabine. The study will last 30 months, from March 1, 2022 to August 30, 2024. The study will be conducted in two reference centers for oncology treatment in the city of Rio de Janeiro.

ELIGIBILITY:
Inclusion Criteria:

* Patients initiating treatment with capecitabine, either: as monotherapy, or in combination with other antineoplastic therapies and/or radiotherapy.
* No restrictions regarding therapeutic regimen or disease stage.
* Age 18 years or older.
* Patients being followed at one or both of the following institutions: Hospital do Câncer I of the National Cancer Institute (INCA), and/or Clementino Fraga Filho University Hospital (UFRJ).

Exclusion Criteria:

* Patients who have previously started capecitabine treatment, with more than one full cycle completed prior to enrollment.
* Inability to communicate verbally or significant difficulty in understanding that prevents adherence to pharmaceutical care instructions.
* Refusal or inability to sign the Informed Consent Form.
* Participation in another clinical study that may interfere with outcomes related to pharmaceutical care.
* Any clinical condition that, in the investigator's judgment, may compromise full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Instruments and questionnaire | Up to 6 months
  Assessment of the clinical benefits of pharmaceutical care, measured by the variation in participants' quality of life between the beginning and end of treatment with capecitabine

SECONDARY OUTCOMES:
Pharmaceutical interventios | Up to 6 months
  Number of pharmaceutical interventions performed

CONTACTS AND LOCATIONS:
Overall Officials: CAMILLE C NIGRI, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; THAISA A NOGUEIRA, PhD, Study Chair — Universidade Federal Fluminense
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
5.204.291
Supporting Information: Study Protocol, CSR
Time Frame: June 2025 - June 2029.
Access Criteria: Results